CLINICAL TRIAL: NCT06402799
Title: Research Protocol for Feasibility Testing of 12 Weeks Home-based E-biking Intervention Among Individuals With Cerebral Palsy
Brief Title: Home-based E-biking Intervention Among Individuals With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-22032100-103168
Record Dates: First submitted 2023-11-03; First posted 2024-05-07 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Palsy
Keywords: Home-based; e-biking; monitoring; cerebral palsy; feasibility
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Feasibility of home-based e-biking among individuals with cerebral palsy. The e-biking intervention consists of 3 sessions per week at the beginning of the study and gradually increases over the training period to 6 sessions per week, with three of these sessions being online and group-supervised.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- E-biking intervention (Experimental): Home-based e-biking
  Interventions: Behavioral: Home-based E-biking

INTERVENTIONS:
Behavioral: Home-based E-biking — The e-biking intervention consists of 3 sessions per week at the beginning of the study and gradually increases over the training period to 6 sessions per week, with three of these sessions being online and group-supervised. Heart rate will be monitored as well as power in Watt at each session.

SUMMARY:
Investigation of the feasibility of virtually group-based e-biking training at home. Individuals aged 13-60 years with CP (Cerebral Palsy) with a Gross Motor Function Classification System score of 1-3 were recruited for a 12-week home-based e-biking training program.

DETAILED DESCRIPTION:
All participants should be able to use a touchscreen, as this type of technology is used in the virtual e-biking training. Participants complete a questionnaire and subsequently engage in 12 weeks of home-based virtual e-biking training. A loaned bicycle will be provided for the training period and set up in the participants' own homes. Setup and adjustments will be performed by trained healthcare personnel. The following measurements will be taken before and after the training period: weight, height, hip-waist measurements, blood pressure, a 30-second sit-to-stand test, a timed-up-and-go test, ankle measurements, and a functional threshold power test (FTP). Seven accelerometers will be attached to the right and left arms, thighs, lower legs, and sternum using NJaP patches and worn for 72 hours at the beginning and end of the training period. The accelerometers can be easily removed after 72 hours.

The e-biking intervention consists of 3 sessions per week at the beginning of the study and gradually increases over the training period to 6 sessions per week, with three of these sessions being online and group-supervised.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with cerebral palsy (GMFCS 1-3)
* Are able to keep balance on a stationary bike
* Are able to use a touchscreen

Exclusion Criteria:

-

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2024-05-18 (Actual)

PRIMARY OUTCOMES:
Feasibility of study assessed by minimum 70% participation in planned training volume among participants | At the end of the study (after 12 weeks of e-biking training)
  Number of participants who complete the study successfully assessed by percentage of completed planned training volume

SECONDARY OUTCOMES:
Change in FTP test among participants | At the end of the study (after 12 weeks of e-biking training)
  The functional threshold power test will change after the intervention as the participants achieve better fitness
Change in timed-up-and-go test | At the end of the study (after 12 weeks of e-biking training)
  The timed-up-an-go test will change after the intervention
Change in the 30-seconds sit-to-stand test | At the end of the study (after 12 weeks of e-biking training)
  The 30-seconds sit-to-stand test will change after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Lorentzen, Professor, Principal Investigator — University of Copenhagen, Department of Neuroscience, Denmark
Locations (1):
- Lisbeth Larsen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No